CLINICAL TRIAL: NCT04473222
Title: Implementing Evidence-based Behavioral Sleep Intervention in Urban Primary Care: Aim 3
Brief Title: Behavioral Sleep Intervention in Urban Primary Care: Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-017788; 5K23HD094905-02 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disturbance; Sleep Deprivation; Sleep
MeSH Terms: conditions — Parasomnias; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Caregiver-child dyads (child ages 1-5 years with a sleep problem) will be recruited from CHOP urban primary care sites and randomly assigned either to the intervention or to an enhanced usual care condition (sleep education handout).
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting outcome assessments will be blinded to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Well! Intervention (Experimental): Participants in this condition will begin the Sleep Well! intervention after initiating baseline, daily diary, and actigraph procedures. Sleep Well! will be provided over approximately 6-8 weeks and will include 3 sessions. Intervention sessions will typically last about an hour, but session length may vary.
  Interventions: Behavioral: Sleep Well!
- Enhanced Usual Care (Other): The enhanced usual care condition will occur between 6 and 8 weeks. At randomization to this condition, participants will be provided with an evidence-based sleep guidelines for young children from the CHOP Parent Family Education manual. Participants in this condition will also be able to consult with their primary care physician for management of child sleep. Consistent with usual care in the CHOP system, the primary care physician may manage the sleep concern or choose to make a referral to the CHOP sleep center or to other behavioral health services internal or external to the CHOP system. Of note, the CHOP Parent Family Education handouts provide contact information for the CHOP Sleep Center and direct readers to follow-up with their primary care provider for further guidance.
  Interventions: Behavioral: Sleep education

INTERVENTIONS:
Behavioral: Sleep Well! — Sleep Well! is a brief, behavioral sleep intervention. The intervention was originally comprised of healthy sleep advice and tested in the context of a sleep health education campaign for impoverished children. Based on preliminary research regarding the need for sleep intervention in primary care, Investigators have expanded the intervention to more comprehensively address poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers who are living in disadvantaged contexts. Intervention components are based on effective pediatric behavioral sleep treatments.
  Arms: Sleep Well! Intervention
Behavioral: Sleep education — Sleep education for caregivers of toddlers and preschoolers is provided via a Parent Family Education handout available to families and clinicians in the CHOP primary care network. The handout contains evidence-based advice about healthy sleep in early childhood.
  Arms: Enhanced Usual Care

SUMMARY:
Investigators will enroll up to 120 parent-child dyads from Children's Hospital of Philadelphia (CHOP) urban primary care clinics. The primary objective of this randomized clinical trial is to determine the whether the Sleep Well! behavioral sleep intervention is feasible and acceptable to families. The investigators will also examine the direction and magnitude in any change in child sleep and child behavior.

DETAILED DESCRIPTION:
Behavioral sleep problems such as insomnia and insufficient sleep are common in toddlers and preschoolers and disproportionately impact lower socioeconomic status (SES) children. Despite a robust evidence base, behavioral sleep interventions are rarely tested with lower-SES children or in primary care, an accessible service delivery setting. The primary objective of this study is to determine whether the Sleep Well! behavioral sleep intervention is feasible and acceptable to families. The investigators will also examine the direction and magnitude of change in child sleep and behavior from pre-intervention to post-intervention and follow-up. This is a randomized controlled trial of the Sleep Well! program with pre-intervention, post-intervention, and follow-up assessments. Caregiver-child dyads (child ages 1-5 years with a sleep problem) will be recruited from CHOP urban primary care sites.

Sleep Well! is a brief, behavioral sleep intervention for toddlers and preschoolers who have a caregiver-reported behavioral sleep problem or who are not getting enough sleep. The intervention includes evidence-based behavioral sleep approaches and strategies to engage and empower families. The primary outcomes for this pilot trial are feasibility (number of caregivers recruited, engaged, and retained in intervention; participant intervention attendance rate) and caregiver acceptability, assessed via a questionnaire and qualitative post-intervention interview. Secondary outcomes are the direction and magnitude in any change in child sleep. Tertiary outcomes are the direction and magnitude in change in child behavior. Assessments occur at pre-intervention, post-intervention, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Parental/guardian permission (informed consent)
2. Caregiver participant is the parent or legal guardian of the child subject
3. Caregiver/legal guardian is greater than or equal to 18 years of age.
4. Child between the ages of 1 and 5 years.
5. Presence of caregiver-reported child sleep problem determined by a Brief Child Sleep Questionnaire item included in an eligibility screening questionnaire or child meets American Academy of Sleep Medicine diagnostic criteria for either pediatric insomnia or insufficient sleep, assessed through an eligibility screening questionnaire.
6. English-speaking.

Exclusion Criteria:

1. Caregiver is not parent or legal guardian of child participant.
2. Presence of a child neurodevelopmental (e.g., autism spectrum disorder; Trisomy 21) or chronic medical (e.g., sickle cell disease, cancer) concern in which the disorder or treatment of the disorder impact sleep.
3. Caregivers/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Williamson, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meltzer LJ, Mindell JA. Systematic review and meta-analysis of behavioral interventions for pediatric insomnia. J Pediatr Psychol. 2014 Sep;39(8):932-48. doi: 10.1093/jpepsy/jsu041. Epub 2014 Jun 19. PMID 24947271
- [Background] Mindell JA, Williamson AA. Benefits of a bedtime routine in young children: Sleep, development, and beyond. Sleep Med Rev. 2018 Aug;40:93-108. doi: 10.1016/j.smrv.2017.10.007. Epub 2017 Nov 6. PMID 29195725
- [Background] Quach J, Gold L, Arnup S, Sia KL, Wake M, Hiscock H. Sleep well--be well study: improving school transition by improving child sleep: a translational randomised trial. BMJ Open. 2013 Oct 28;3(10):e004009. doi: 10.1136/bmjopen-2013-004009. PMID 24165031
- [Background] Allen SL, Howlett MD, Coulombe JA, Corkum PV. ABCs of SLEEPING: A review of the evidence behind pediatric sleep practice recommendations. Sleep Med Rev. 2016 Oct;29:1-14. doi: 10.1016/j.smrv.2015.08.006. Epub 2015 Sep 1. PMID 26551999
- [Background] Williamson AA, Milaniak I, Watson B, Cicalese O, Fiks AG, Power TJ, Barg FK, Beidas RS, Mindell JA, Rendle KA. Early Childhood Sleep Intervention in Urban Primary Care: Caregiver and Clinician Perspectives. J Pediatr Psychol. 2020 Sep 1;45(8):933-945. doi: 10.1093/jpepsy/jsaa024. PMID 32430496
- [Background] Mindell JA, Sedmak R, Boyle JT, Butler R, Williamson AA. Sleep Well!: A Pilot Study of an Education Campaign to Improve Sleep of Socioeconomically Disadvantaged Children. J Clin Sleep Med. 2016 Dec 15;12(12):1593-1599. doi: 10.5664/jcsm.6338. PMID 27655459
- See also: Created by the Pediatric Sleep Council, babysleep.com provides comprehensive and expert-based information on baby and toddler sleep that is freely available to the public. — http://babysleep.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregiver-child dyads (child ages 1-5 years with a sleep problem) were recruited from pediatrician referrals, chart reviews, and study flyers at 3 urban (i.e., large, metropolitan) primary care sites affiliated with Children's Hospital of Philadelphia (CHOP).
Pre-assignment Details: 104 caregiver-child dyads were randomly assigned to either the intervention group or enhanced usual care group immediately following consent. The number in each group shown reflects dyads and not individual caregivers and/or individual children.
Groups:
- Sleep Well! Intervention: Caregiver-child dyads in this condition will begin the Sleep Well! intervention after initiating baseline, daily diary, and actigraph procedures. Sleep Well! will be provided over approximately 6-8 weeks and will include 3 sessions. Intervention sessions will typically last about an hour, but session length may vary.
  Sleep Well!: Sleep Well! is a brief, behavioral sleep intervention. The intervention was originally comprised of healthy sleep advice and tested in the context of a sleep health education campaign for impoverished children. Based on preliminary research regarding the need for sleep intervention in primary care, Investigators have expanded the intervention to more comprehensively address poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers who are living in disadvantaged contexts. Intervention components are based on effective pediatric behavioral sleep treatments.
- Enhanced Usual Care: The enhanced usual care condition will occur between 6 and 8 weeks. At randomization to this condition, caregiver-child dyads will be provided with an evidence-based sleep guidelines for young children from the CHOP Parent Family Education manual. Caregiver-child dyads in this condition will also be able to consult with their primary care physician for management of child sleep. Consistent with usual care in the CHOP system, the primary care physician may manage the sleep concern or choose to make a referral to the CHOP sleep center or to other behavioral health services internal or external to the CHOP system. Of note, the CHOP Parent Family Education handouts provide contact information for the CHOP Sleep Center and direct readers to follow-up with their primary care provider for further guidance.
  Sleep education: Sleep education for caregivers of toddlers and preschoolers is provided via a Parent Family Education handout available to families and clinicians in the CHOP primary care network. The handout contains evidence-based advice about healthy sleep in early childhood.
Period: Overall Study
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Started | 52 (104 unique participants (52 caregiver-child dyads) started the study. The numbers reflected in the table represent the number of caregiver-child dyads that participated in the study. 2 caregiver-child dyads lost contact after consent and did not initiate baseline measures.) | 52 (104 unique participants (52 caregiver-child dyads) started the study. The numbers reflected in the table represent the number of caregiver-child dyads that participated in the study. 4 caregiver-child dyads lost contact after consenting and did not initiate baseline measures.)
Baseline | 50 | 47 (1 caregiver-child dyad partially completed baseline surveys, then lost contact, then re-contacted and were re-consented as a new caregiver-child dyad with new identification number in this condition.)
Time 2/Post-intervention | 44 (6 caregiver-child dyads lost contact between baseline and time 2 (post-intervention).) | 43 (4 caregiver-child dyads lost contact between baseline and time 2)
Completed | 39 (78 unique participants (39 caregiver-child dyads) completed the study. 4 caregiver-child dyads lost contact between time 2 (post-intervention) and time 3 (follow-up); 1 caregiver-child dyad started but did not complete the time 3 (follow-up) assessment.) | 37 (74 unique participants (37 caregiver-child dyads) completed the study. 3 caregiver-child dyads lost contact between time 2 (post-intervention) and time 3 (follow-up); 1 caregiver-child dyad withdrew while completing the time 3 (follow-up assessment); 2 caregiver-child dyads started but did not complete the time 3 (follow-up) assessment.)
Not Completed | 13 | 15
Not completed — Lost to Follow-up | 13 | 13
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Participant partially completed baseline surveys, then lost contact, then re-consented | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants reflect the total number of children and caregivers in each arm (i.e., 100 participants or 50 caregiver-child dyads in the Sleep Well! intervention, and 94 participants or 47 caregiver-child dyads in enhanced usual care). Because 7 caregivers and 7 children (n=14, or 7 caregiver-child dyads) did not complete baseline, there were N=194 evaluable participants (n=97 children and n=97 caregivers), or 97 evaluable caregiver-child dyads total.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Categorical [Count of Participants; unit: Participants] — Population: This information is for the caregiver participants only in the caregiver-child dyad. Caregivers reported their age by responding to a categorical question with age group brackets.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 50 | 47 | 97
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This information is for the child participants in the caregiver-child dyad. Age in years for the participating child was drawn from their medical record.
  years
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 2.50 (1.18) | 2.55 (1.32) | 2.52 (1.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This information is for the child participants in the caregiver-child dyad. The participating child's sex at birth was drawn from their medical record.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Female | 20 | 25 | 45
    Male | 30 | 22 | 52
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This information is for the caregiver participants in the caregiver-child dyad. Caregivers reported their sex by responding to categorical survey question.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Female | 48 | 46 | 94
    Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the child participants in the caregiver-child dyad. The participating child's race and ethnicity were drawn from their medical record.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Hispanic or Latino | 2 | 6 | 8
    Not Hispanic or Latino | 48 | 41 | 89
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the caregiver participants in the caregiver-child dyad. Caregivers responded to a categorical item to report their ethnic background.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Hispanic or Latino | 2 | 4 | 6
    Not Hispanic or Latino | 48 | 43 | 91
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the child participants in the caregiver-child dyad. The participating child's race and ethnicity were drawn from their medical record.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 33 | 36 | 69
    White | 10 | 10 | 20
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This information is for the caregiver participants in the caregiver-child dyad. Caregivers responded to a categorical item to report their racial background.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 32 | 35 | 67
    White | 12 | 8 | 20
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants] — This information reflects both members of the caregiver-child dyad (50 children and 50 caregivers in Sleep Well! arm [total = 100], 47 children and 47 caregivers in enhanced usual care arm [total = 94]). Region of enrollment was drawn from study records documenting the location of the primary care site from which the participants were recruited.
  participants
    United States | 100 | 94 | 194
Caregiver educational attainment [Count of Participants; unit: Participants] — Population: This information is for the caregiver participants in the caregiver-child dyad. Caregivers reported on their highest level of educational attainment, which was dichotomized to reflect education of high school or less and education of more than high school.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Greater than high school education | 30 | 32 | 62
    High school education or less | 20 | 15 | 35
Family living at or below 125% of the US poverty line [Count of Participants; unit: Participants] — Population: This information reflects the caregiver within the caregiver-child dyad. Caregivers reported on their family size and household income, which were used to determine whether families were living at 125% or below the US federal poverty line, according to US guidelines.
  Participants
    number analyzed (Participants) | 50 | 47 | 97
    Living at or below 125% of the poverty line | 22 | 17 | 39
    Living above 125% of the poverty line | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate (Intervention Feasibility)
Description: The study team will track the number of caregiver-child dyad participants assigned to the Sleep Well! condition who complete the intervention as a measure of retention, or intervention feasibility. The retention rate reported is for those who completed all sessions and phone calls for the Sleep Well! intervention.
Time Frame: Study duration (up to 24 weeks)
Population: Percentage of caregiver-child dyads that completed all sessions of Sleep Well! of those who initiated the intervention. Results for this outcome are not reported for the Enhanced Usual Care condition, as this outcome pertains only to those who initiated the Sleep Well! intervention. This is a descriptive outcome, and no statistical comparisons were conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention
Number analyzed (Participants) | 50
Participants
  Completed all 3 sessions and all 3 phone calls | 46
  Did not complete all 3 sessions and/or all 3 phone calls | 4

2. Primary Outcome: Family Engagement (Sessions)
Description: For families randomized to the intervention condition, study interventionists will rate family engagement during telehealth sessions using a one-item 5-point Likert scale ranging from 1 (not engaged) to 5 (very good engagement), with higher scores representing better engagement. The outcome reported is the average rating of telehealth session engagement across sessions 1, 2, and 3.
Time Frame: Study duration (up to 24 weeks)
Population: The analytic sample is based on the 49 caregiver-child dyads that attended at least 1 session. Of the 50 dyads that completed baseline measures, 1 dyad lost contact prior to the start of intervention and thus is not included. Results are not reported for the Enhanced Usual Care dyads, as this outcome pertains only to those who initiated the Sleep Well! intervention. This is a descriptive outcome without any statistical comparisons.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sleep Well! Intervention: Participants in this condition will begin the Sleep Well! intervention after initiating baseline, daily diary, and actigraph procedures. Sleep Well! will be provided over approximately 6-8 weeks and will include 3 sessions and 3 follow-up phone calls. Intervention sessions will typically last about an hour, but session length may vary.
  Sleep Well!: Sleep Well! is a brief, behavioral sleep intervention. The intervention was originally comprised of healthy sleep advice and tested in the context of a sleep health education campaign for impoverished children. Based on preliminary research regarding the need for sleep intervention in primary care, Investigators have expanded the intervention to more comprehensively address poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers who are living in disadvantaged contexts. Intervention components are based on effective pediatric behavioral sleep treatments.
Arm/Group | Sleep Well! Intervention
Number analyzed (Participants) | 49
units on a scale | 4.58 (0.66)

3. Primary Outcome: Family Engagement (Telephone Calls)
Description: For families randomized to the intervention condition, study interventionists will rate family engagement during telephone calls using a one-item 5-point Likert scale ranging from 1 (not engaged) to 5 (very good engagement), with higher scores representing better engagement. The outcome reported is the average rating of telehealth session engagement across all completed telephone calls.
Time Frame: Study duration (up to 24 weeks)
Population: The analytic sample is based on the 49 caregiver-child dyads that completed at least 1 telephone call. Of the 50 dyads that completed baseline measures, 1 dyad lost contact prior to the start of intervention and thus is not included. Results are not reported for the Enhanced Usual Care dyads, as this outcome pertains only to those who initiated the Sleep Well! intervention. This is a descriptive outcome without any statistical comparisons.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sleep Well! Intervention
Number analyzed (Participants) | 49
units on a scale | 4.59 (0.66)

4. Primary Outcome: Treatment Acceptability
Description: Caregivers will complete the Treatment Evaluation Inventory-Short Form, a widely used measure of treatment acceptability that has been adapted for the purposes of the Sleep Well! intervention. For this reported outcome, caregivers responded to the statement "I found these strategies to be an acceptable way of dealing with my child's sleep" on a 5-point Likert scale ranging from 1 "strongly disagree" to 5 "strongly agree," with higher scores reflecting stronger acceptability.
Time Frame: Time 2 (an average of 9 weeks post-baseline)
Population: The analytic sample is based on the 44 intervention participants that completed Sleep Well! and time 2 (post-intervention) surveys. Of the 50 that completed baseline, 1 lost contact prior to attending any sessions, 3 lost contact during intervention, and 2 lost contact after the intervention but before post-intervention. Results are not reported for Enhanced Usual Care, as this outcome pertains to the Sleep Well! intervention. This is a descriptive outcome without any statistical comparisons.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention
Number analyzed (Participants) | 44
Participants
  Strongly agree | 28
  Agree | 13
  Neutral | 2
  Disagree | 0
  Strongly disagree | 1

5. Primary Outcome: Treatment Acceptability: Cultural Humility
Description: Caregivers will complete the Multicultural Therapy Competency Inventory- Client Version, adapted for the current study, to assess participants' perceptions of the Sleep Well! therapist's cultural humility during the intervention. Caregivers in the intervention condition responded to the statement "When we discussed my child's sleep, my Sleep Well! therapist was accepting of my family's values and beliefs," on a 5-point Likert scale ranging from 1 "strongly disagree" to 5 "strongly agree." Higher ratings indicate greater perceived cultural humility.
Time Frame: Time 2 (an average of 9 weeks post-baseline)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention
Number analyzed (Participants) | 44
Participants
  Strongly agree | 36
  Agree | 4
  Neutral | 1
  Disagree | 0
  Strongly disagree | 3

6. Primary Outcome: Assessment Process (Study Feasibility)
Description: The study team will keep records of the number of planned assessments that are completed (i.e., the entire assessment was completed) as a measure of study feasibility.
Time Frame: Study duration (up to 24 weeks)
Population: The analytic sample was based on the participants that completed baseline measures (50 Sleep Well! and 47 Enhanced Usual Care participants). This is a descriptive outcome and no statistical comparisons were made.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Participants
  Baseline (pre-intervention) | 50 | 47
  Time 2 (an average of 9 weeks post-baseline) | 44 | 43
  Time 3 (an average of 15 weeks post-baseline) | 39 | 37

7. Secondary Outcome: Severity of Child Sleep Problems
Description: Caregivers will complete a Brief Child Sleep Questionnaire item to report on the severity of any caregiver-perceived sleep problems at pre-intervention, post-intervention, and follow-up. Caregivers reported on the severity of child sleep problems on a 5-point Likert scale; responses were then dichotomized as in prior research such that 0= no to very small sleep problem and 1= small, moderate, or serious sleep problem. Higher scores indicate worse sleep problems.
Time Frame: Baseline (pre-intervention), Time 2 (an average of 9 weeks post-baseline), and Time 3 (an average of 15 weeks post-baseline)
Population: Analysis was based on the sample that completed baseline (pre-intervention) measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Participants
  Baseline (pre-intervention) | 45 | 38
  Time 2 (an average of 9 weeks post-baseline) | 20 | 33
  Time 3 (an average of 15 weeks post-baseline) | 13 | 21
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = .026, t-test, 2 sided; Odds Ratio, log = -0.15 — The logit represents the difference in log odds per 1-week change in time for the intervention group relative to enhanced usual care

8. Secondary Outcome: Child Sleep Problems: Bedtime Difficulties
Description: Caregivers will complete a Brief Child Sleep Questionnaire item to report on the severity of child bedtime difficulties at pre-intervention, post-intervention, and follow-up. Caregivers reported on the severity of bedtime difficulties on a 5-point Likert scale; responses were then dichotomized as in prior research such that 0= easy to somewhat easy bedtime and 1= somewhat difficult, difficult, or very difficult at bedtime. Higher scores indicate greater bedtime difficulties.
Time Frame: as for outcome 7
Population: Analysis was based on the sample that completed baseline (pre-intervention) measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Participants
  Baseline (pre-intervention) | 41 | 36
  Time 2 (an average of 9 weeks post-baseline) | 18 | 30
  Time 3 (an average of 15 weeks post-baseline) | 14 | 22
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.032, t-test, 2 sided; Odds Ratio, log = -0.20 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Child Sleep Patterns: Sleep Onset Latency
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits (sleep time, total sleep duration, night wakings, aspects of the sleep environment, etc.) at pre-intervention, post-intervention, and follow-up. The BCSQ is appropriate for children ages 1-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. Caregivers responded to a BCSQ question regarding the time the child took to fall asleep in minutes after lights out. Higher values indicate a longer period of time to fall asleep in minutes.
Time Frame: as for outcome 7
Population: The analytic sample is based on participants that completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Minutes
  Baseline (pre-intervention) | 57.00 (46.24) | 52.34 (36.70)
  Time 2 (an average of 9 weeks post-baseline) | 31.02 (35.35) | 42.79 (35.78)
  Time 3 (an average of 15 weeks post-baseline) | 29.13 (31.09) | 38.08 (32.56)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = .010, t-test, 2 sided; Slope = -0.01, Standard Error of Mean .009 — The estimate represents the differential change in slope per week for the intervention group relative to enhanced usual care

10. Secondary Outcome: Child Sleep Patterns: Number of Wakings Per Night
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits (sleep time, total sleep duration, night wakings, aspects of the sleep environment, etc.) at pre-intervention, post-intervention, and follow-up. The BCSQ is appropriate for children ages 1-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. Caregivers responded to a BCSQ question regarding the number of times their child woke during the night. Higher values indicate more frequent wakings per night.
Time Frame: as for outcome 7
Population: The analytic sample is based on participants that completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Wakings
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Wakings
  Baseline (pre-intervention) | 1.84 (1.54) | 1.85 (1.16)
  Time 2 (an average of 9 weeks post-baseline) | 1.27 (1.07) | 1.37 (1.11)
  Time 3 (an average of 15 weeks post-baseline) | 1.02 (1.12) | 1.23 (1.06)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.161, t-test, 2 sided; Slope = 0.009, Standard Error of Mean 0.009 — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Child Sleep Patterns: Duration of Wakings Per Night
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits (sleep time, total sleep duration, night wakings, aspects of the sleep environment, etc.) at pre-intervention, post-intervention, and follow-up. The BCSQ is appropriate for children ages 1-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. Caregivers responded to a BCSQ question regarding the total time in minutes their child was awake during the night. Higher values indicate longer night wakings in minutes.
Time Frame: as for outcome 7
Population: The analytic sample is based on participants that completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Minutes
  Baseline (pre-intervention) | 106.80 (162.48) | 71.81 (113.85)
  Time 2 (an average of 9 weeks post-baseline) | 58.64 (109.07) | 78.49 (132.51)
  Time 3 (an average of 15 weeks post-baseline) | 21.38 (38.11) | 89.62 (175.08)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.006, t-test, 2 sided; Slope = -0.03, Standard Error of Mean 0.01 — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Child Sleep Patterns: Nighttime Sleep Duration
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits (sleep time, total sleep duration, night wakings, aspects of the sleep environment, etc.) at pre-intervention, post-intervention, and follow-up. The BCSQ is appropriate for children ages 1-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. Caregivers responded to a BCSQ question regarding the total time their child slept overnight in hours. Higher values indicate longer nighttime sleep duration in hours.
Time Frame: as for outcome 7
Population: The analytic sample is based on participants that completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Hours
  Baseline (pre-intervention) | 7.58 (2.46) | 7.99 (2.62)
  Time 2 (an average of 9 weeks post-baseline) | 8.73 (1.86) | 8.39 (2.06)
  Time 3 (an average of 15 weeks post-baseline) | 8.73 (2.11) | 8.19 (2.07)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.045, t-test, 2 sided; Slope = 0.07, Standard Error of Mean 0.04 — [estimate comment as in outcome 9, analysis 1]

13. Secondary Outcome: Child Sleep Patterns: Total 24-hour Sleep Duration
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits (sleep time, total sleep duration, night wakings, aspects of the sleep environment, etc.) at pre-intervention, post-intervention, and follow-up. The BCSQ is appropriate for children ages 1-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. Caregivers responded to a BCSQ question regarding the total time their child slept overnight, and a BCSQ question regarding the total time their child slept during the day for naps. Responses to these two items were summed to estimate total (24-hour) sleep duration in hours. Higher values indicate longer total sleep duration in hours.
Time Frame: as for outcome 7
Population: The analytic sample is based on participants that completed the baseline assessment.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
Hours
  Baseline (pre-intervention) | 9.53 (3.40) | 9.88 (3.48)
  Time 2 (an average of 9 weeks post-baseline) | 10.61 (2.81) | 10.18 (2.68)
  Time 3 (an average of 15 weeks post-baseline) | 10.29 (2.42) | 10.07 (2.88)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.685, t-test, 2 sided; Slope = -0.05, Standard Error of Mean 0.11 — [estimate comment as in outcome 9, analysis 1]

14. Secondary Outcome: Child Sleep Patterns: Actigraphy Derived Nighttime Sleep Duration
Description: Caregivers will have their child wear an actigraph to obtain estimates of sleep onset, sleep offset, and sleep duration at pre-intervention, post-intervention, and follow-up. Nighttime sleep duration in minutes is obtained from scoring sleep onset and sleep offset in combination with caregiver-reported nightly sleep diaries of bed and wake times. Nighttime sleep duration is expressed as the average sleep duration in minutes across the 7 nights of actigraphy at each timepoint. Higher values indicate longer average nighttime sleep duration.
Time Frame: 7 days at Baseline (pre-intervention), Time 2 (an average of 9 weeks post-baseline), and Time 3 (an average of 15 weeks post-baseline)
Population: Analytic sample was based on the number of participants that completed actigraphy. Of the 50 intervention participants that initiated baseline, 11 did not complete actigraphy assessment due to losing contact or opting out of this assessment procedure. Of the 47 enhanced usual care participants that initiated baseline, 9 did not complete actigraphy assessment due to losing contact or opting out of this assessment procedure.
Measure: Mean (Standard Deviation); unit: Minutes per night
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 39 | 38
Minutes per night
  Baseline (pre-intervention) | 556.97 (51.78) | 559.96 (58.08)
  Time 2 (an average of 9 weeks post-baseline) | 545.45 (84.24) | 554.29 (76.57)
  Time 3 (an average of 15 weeks post-baseline) | 571.40 (72.26) | 557.69 (60.97)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.734, t-test, 2 sided; Slope = 0.42, Standard Error of Mean 1.22 — [estimate comment as in outcome 9, analysis 1]

15. Secondary Outcome: Child Behavior Problems: Externalizing Problems
Description: Caregivers will complete the Child Behavioral Checklist (CBCL) for ages 1.5-5 years to report on child internalizing and externalizing concerns at Baseline, Time 2 (post-intervention), and Time 3 (follow-up). The CBCL has shown strong reliability and validity in large validation studies and is a widely used measure of child behavior. The Externalizing T-score is generated from caregiver-rated raw items that are summed and converted to T-scores based on CBCL normative data. Higher T-scores indicate greater externalizing problems. 50 indicates the population mean with a standard deviation of 10. A T-score of 65-69.9 indicates elevated concerns and a T-score of 70 and above indicates clinically significant concerns.
Time Frame: as for outcome 7
Population: The analytic sample was based on the participants that completed baseline measures.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
T-score
  Baseline (pre-intervention) | 50.32 (11.45) | 45.68 (11.43)
  Time 2 (an average of 9 weeks post-baseline) | 46.41 (12.09) | 44.14 (11.54)
  Time 3 (an average of 15 weeks post-baseline) | 44.84 (10.85) | 44.47 (11.52)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.019, t-test, 2 sided; Slope = -0.20, Standard Error of Mean 0.08 — [estimate comment as in outcome 9, analysis 1]

16. Secondary Outcome: Child Behavior Problems: Internalizing Problems
Description: Caregivers will complete the Child Behavioral Checklist (CBCL) for ages 1.5-5 years to report on child internalizing and externalizing concerns at Baseline, Time 2 (post-intervention), and Time 3 (follow-up). The CBCL has shown strong reliability and validity in large validation studies and is a widely used measure of child behavior. The Internalizing T-score is generated from caregiver-rated raw items that are summed and converted to T-scores based on CBCL normative data. Higher T-scores indicate greater internalizing problems. 50 indicates the population mean with a standard deviation of 10. A T-score of 65-69.9 indicates elevated concerns and a T-score of 70 and above indicates clinically significant concerns.
Time Frame: as for outcome 7
Population: The analytic sample was based on the participants that completed baseline measures.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Sleep Well! Intervention | Enhanced Usual Care
Number analyzed (Participants) | 50 | 47
T-score
  Baseline | 47.39 (10.54) | 43.20 (10.23)
  Time 2 (an average of 9 weeks post-baseline) | 44.20 (9.49) | 43.05 (12.46)
  Time 3 (an average of 15 weeks post-baseline) | 44.54 (11.19) | 41.37 (10.86)
Statistical Analysis 1: Comparison: Sleep Well! Intervention vs Enhanced Usual Care; Test type: Superiority; p = 0.776, t-test, 2 sided; Slope = -0.04, Standard Error of Mean 0.14 — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored by the study team throughout each participating caregiver-child dyad's study participation, which was up to 24 weeks.
Description: This was a minimal risk behavioral intervention for a child sample and as such, serious adverse events and all-cause mortality risks were not expected.
Groups:
- Sleep Well! Intervention Child Participants; Sleep Well! Intervention Caregiver Participants: Caregiver-child dyads in this condition will begin the Sleep Well! intervention after initiating baseline, daily diary, and actigraph procedures. Sleep Well! will be provided over approximately 6-8 weeks and will include 3 sessions. Intervention sessions will typically last about an hour, but session length may vary.
  Sleep Well!: Sleep Well! is a brief, behavioral sleep intervention. The intervention was originally comprised of healthy sleep advice and tested in the context of a sleep health education campaign for impoverished children. Based on preliminary research regarding the need for sleep intervention in primary care, Investigators have expanded the intervention to more comprehensively address poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers who are living in disadvantaged contexts. Intervention components are based on effective pediatric behavioral sleep treatments.
- Enhanced Usual Care Child Participants; Enhanced Usual Care Caregiver Participants: The enhanced usual care condition will occur between 6 and 8 weeks. At randomization to this condition, caregiver-child dyads will be provided with an evidence-based sleep guidelines for young children from the CHOP Parent Family Education manual. Caregiver-child dyads in this condition will also be able to consult with their primary care physician for management of child sleep. Consistent with usual care in the CHOP system, the primary care physician may manage the sleep concern or choose to make a referral to the CHOP sleep center or to other behavioral health services internal or external to the CHOP system. Of note, the CHOP Parent Family Education handouts provide contact information for the CHOP Sleep Center and direct readers to follow-up with their primary care provider for further guidance.
  Sleep education: Sleep education for caregivers of toddlers and preschoolers is provided via a Parent Family Education handout available to families and clinicians in the CHOP primary care network. The handout contains evidence-based advice about healthy sleep in early childhood.
Arm/Group | Sleep Well! Intervention Child Participants | Enhanced Usual Care Child Participants | Sleep Well! Intervention Caregiver Participants | Enhanced Usual Care Caregiver Participants
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47 | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47 | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47 | 0/50 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04473222/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04473222/ICF_001.pdf